CLINICAL TRIAL: NCT04530513
Title: ARREST - A Phase I Study of SABR for Poly-metastatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Glenn Bauman, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARREST; ReDA #10401 (Other: Lawson Health Research Institute)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancer
Keywords: Stereotatic ablative radiotherapy; Poly-Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Dose Escalation Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose Level 1 (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy - Level 1
- Dose Level 2 (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy - Level 2
- Dose Level 3 (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy - Level 3
- Dose Level 4 (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy - Level 4
- De-escalation Level (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy - De-escalation Level

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy - Level 1 — 6Gy x 2 fractions to all sites in 2 weeks
  Arms: Dose Level 1
Radiation: Stereotactic ablative radiotherapy - Level 2 — 6Gy x 3 fractions to all sites in 3 weeks
  Arms: Dose Level 2
Radiation: Stereotactic ablative radiotherapy - Level 3 — 6Gy x 4 fractions to all sites in 4 weeks
  Arms: Dose Level 3
Radiation: Stereotactic ablative radiotherapy - Level 4 — 6Gy x 5 fractions to all sites in 5 weeks
  Arms: Dose Level 4
Radiation: Stereotactic ablative radiotherapy - De-escalation Level — 6Gy x 1 fraction to all sites in 1 week
  Arms: De-escalation Level

SUMMARY:
Stereotactic ablative radiotherapy (SABR) is a new radiation treatment that delivers high-dose, precise radiation to small areas in the body. This new technique can potentially allow radiation treatments to be focused more precisely, and be delivered more accurately than with older treatments. This improvement could help by reducing side effects overall (through radiation exposure to a smaller area of the body over a shorter time period), and by improving the chance of controlling the cancer by more precisely treating the cancer and by giving higher doses of radiation. SABR is considered a standard treatment for some lung cancers, and selected cancers that have spread to the brain. Ongoing studies are evaluating the use of SABR for treating people with up to 10 sites of cancer in the body, but its safety and value for treating patients with poly-metastatic cancer (more than 10 sites of cancer) is not yet known.

The purpose of this study is to determine the safety of using SABR to treat people with poly-metastatic disease. To our knowledge, this is the first time that SABR will be tested in people who have poly-metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to provide informed consent
* ECOG 0-2
* Life expectancy greater than 3 months
* Histologically confirmed malignancy with metastatic disease detected on imaging. A biopsy of a metastatic site is preferred, but not required.
* Staging/Re-staging within 6 weeks prior to enrollment:

  * Brain: Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) for tumor sites with propensity for brain metastasis. All patients with brain metastases (at enrollment or previously treated) require an MRI of the brain.
  * Body: CT neck/chest/abdomen/pelvis and bone scan required. This may be replaced with a Positron Emission Tomography (PET)/CT (18-Fluorodeoxyglucose [FDG] or Prostate Specific Membrane Antigen [PSMA]) except for tumors where FDG uptake is not expected.
  * Spine: MRI of the spine is not mandatory for enrollment.
* Presence of poly-metastatic disease, defined as total number of targets greater than 10
* No standard of care systemic therapy option exists for the patient, the patient refuses further standard systemic therapy, or there is no intent to deliver systemic therapy for 3 months after enrollment.
* At the discretion of the treating oncologist, it is believed that all sites of disease can be safely treated for enrollment on study.

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy. These include interstitial lung disease in patients requiring thoracic radiation, Crohn's disease in patients where the Gastrointestinal (GI) tract will receive radiotherapy, ulcerative colitis where the bowel will receive radiotherapy or connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction
* Inadequate baseline bone marrow function (i.e. symptomatic anemia, neutropenia and/or thrombocytopenia which may interfere with the ability to deliver radiation).
* Chronic kidney dysfunction Estimated Glomerular Filtration Rate (eGFR) less than 30 where a significant dose of radiotherapy is expected to be delivered to the kidney.
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses.
* Prior treatment with systemic radiopharmaceuticals (i.e. Radium 223 or Lutetium 177)
* More than 50 metastases (count excluding equivocal lesions less than 5mm in size)
* Any single metastasis greater than 5 cm in size. This is a firm cut-off.
* Any brain metastasis greater than 3 cm in size or a total volume of brain metastases greater than 30 cc. This is a firm cut-off.
* Central Nervous System (CNS) only disease
* Metastasis in the brainstem.
* Inability to treat all sites of disease, which may include:

  * Disease involving any of the following: GI tract (including esophagus, stomach, small or large bowel), mesenteric lymph nodes, and/or skin
  * Diffuse or "miliary" metastatic disease of brain, bone, lung, liver or other sites (i.e. lymphangitic spread, malignant pleural effusion/ascites, peritoneal disease, leptomeningeal metastases) where it would be impossible to deliver radiotherapy at the intended dose level
* Any evidence of epidural disease on any baseline imaging.
* Clinical or radiologic evidence of spinal cord compression.
* Dominant brain metastasis requiring surgical decompression.
* Patients treated with prior systemic therapy are eligible for this study, however, systemic therapy agents that are cytotoxic, immunotherapeutic, or molecularly targeted agents are NOT allowed within the period of time commencing 2 weeks prior to radiation. Patients on conventional hormone therapy with anti-estrogen therapy (including but not limited to tamoxifen, letrozole, anastrozole, Luteinizing Hormone-Releasing Hormone [LHRH] agonists or antagonists) or anti-testosterone therapy (including but not limited to LHRH agonists or antagonists, direct anti-androgens like bicalutamide, apalutamide or steroid synthesis inhibitors like abiraterone) may continue this medication. No systemic therapy may be planned to initiate within 6 weeks after completion of radiotherapy.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose of Stereotactic Radiotherapy | 2 years and 3 months
  In determining the maximally tolerated dose (MTD) grade 5 toxicity (patient death) attributable to treatment, any Grade 4 toxicity among the Hematologic, Hepatobiliary or Respiratory domains, more than 3 instances of Grade 3-4 toxicities occurring within 6 weeks of treatment will be taken into consideration. This is based on the Common Terminology Criteria for Adverse Events (CTCAE) grading system. Additionally, in determining the MTD, the feasibility of successfully planning and treating at a given dose level will be considered.

SECONDARY OUTCOMES:
Quality of life at 6 weeks post radiotherapy as measured by the Functional Assessment of Cancer Therapy - General (FACT-G) | 2 years and 3 months
  The Functional Assessment of Cancer Therapy - General (FACT-G ) is a standardized questionnaire used to measure quality of life. The questionnaire consists of 4 scales measuring 27 items in total. Categories of the 4 scales are: physical well-being, social/family well-being, emotional well-being, and functional well-being. The score for each item in the scale ranges from 0 to 4, where 0 is not at all and 4 is very much. The scores from each scale are added up, and can be combined to provide a total score.
Quality of life at 6 weeks post radiotherapy as measured by the EuroQOL Group EQ-5D-5L | 2 years and 3 months
  The EQ-5D-5L is a standardized questionnaire used to measure quality of life and health. The first section includes 5 categories: mobility, self-care, usual activities (e.g. work, family), pain/discomfort, and anxiety/depression. Each category contains 5 statements ranging from no problems to extreme problems, where no problems is assigned a code of 1 and extreme problems is assigned a code of 5. Participants are asked to select the statement that best describes their health that day. No score is generated, rather a 5 digit code is generated based on the response provided, which can then be combined into a data set and interpreted in a variety of ways. The second section includes a 20 cm analogue scale from 0 to 100, where 100 is the best health ever imagined and 0 is the worst health imagined. The participant will mark a score on the scale representing the state of their health on that day.
Progression free survival post radiotherapy | 4 years
  Time from randomization to disease progression at any site or death.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute
Locations (1):
- London Health Sciences Centre - London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corkum MT, Fakir H, Palma DA, Nguyen T, Bauman GS. Can Polymetastatic Disease Be ARRESTed Using SABR? A Dosimetric Feasibility Study to Inform Development of a Phase 1 Trial. Adv Radiat Oncol. 2021 Jun 5;6(5):100734. doi: 10.1016/j.adro.2021.100734. eCollection 2021 Sep-Oct. PMID 34278053
- [Derived] Bauman GS, Corkum MT, Fakir H, Nguyen TK, Palma DA. Ablative radiation therapy to restrain everything safely treatable (ARREST): study protocol for a phase I trial treating polymetastatic cancer with stereotactic radiotherapy. BMC Cancer. 2021 Apr 14;21(1):405. doi: 10.1186/s12885-021-08020-2. PMID 33853550